CLINICAL TRIAL: NCT05551910
Title: Comparison of Analgesic and Sedative Effects of Esmketamine and Remifentanil Combined With Propofol Respectively in Septic Shock Patients With Invasive Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Yuting Li, Principal Investigator, The First Hospital of Jilin University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Yuting Li
Record Dates: First submitted 2022-09-08; First posted 2022-09-23 (Actual); Last update posted 2022-09-23 (Actual); Status verified 2022-09

CONDITIONS: Patients With Septic Shock Admitted to the ICU on Invasive Mechanical Ventilation
Keywords: septic shock; invasive mechanical ventilation;ICU
MeSH Terms: conditions — Shock, Septic | interventions — Esketamine; Remifentanil; Propofol

STUDY DESIGN:
Intervention Model Description: RCT
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Analgesia and sedation with esmketamine combined with propofol (Experimental)
  Interventions: Drug: Esketamine; Drug: propofol
- Remifentanil combined with propofol for analgesia and sedation (Other)
  Interventions: Drug: Remifentanil; Drug: propofol

INTERVENTIONS:
Drug: Esketamine — The patients in the test group were given esmketamine (50mg / 2ml * branch, Jiangsu Hengrui Pharmaceutical Co., Ltd.) 0.15-0.5mg/kg H was pumped intravenously. Two minutes after the administration, the pain was scored with the cpot pain observation scale. The target cpot was < 3 points. The dose of esketamine was adjusted according to the cpot score.
  Arms: Analgesia and sedation with esmketamine combined with propofol
Drug: Remifentanil — Patients in the control group were given remifentanil (1mg / branch, Yichang humanwell Pharmaceutical Co., Ltd.) 0.05-2ug/kg Minutes after administration, the analgesic score was measured with cpot pain observation scale. The target cpot was less than 3 points, and the dose of remifentanil was adjusted according to the cpot score.
  Arms: Remifentanil combined with propofol for analgesia and sedation
Drug: propofol — propofol

SUMMARY:
Septic shock patients with invasive mechanical ventilation who were randomly enrolled in ICU were divided into esketamine group (test group) and remifentanil group (control group) according to the ratio of 1:1. The dose of vasopressor, the time of mechanical ventilation, the incidence of intestinal dysfunction and the dose of propofol were compared between the two groups. Through statistical analysis, it was determined whether esketamine combined with propofol could improve the prognosis of septic shock patients with invasive mechanical ventilation and reduce the adverse reactions of analgesic and sedative drugs compared with remifentanil combined with propofol.

DETAILED DESCRIPTION:
The purpose of this study is to determine whether esketamine combined with propofol can improve the prognosis and reduce the adverse effects of analgesic and sedative drugs in septic shock patients undergoing invasive mechanical ventilation compared with remifentanil combined with propofol.

Study methods: septic shock patients with invasive mechanical ventilation in ICU were randomly divided into esketamine group (test group) and remifentanil group (control group) according to the ratio of 1:1. 120 patients are expected to be enrolled. The dose of vasopressor, the time of mechanical ventilation, the incidence of intestinal dysfunction and the dose of propofol were compared between the two groups. Through statistical analysis, it was determined whether esketamine combined with propofol could improve the prognosis of septic shock patients with invasive mechanical ventilation and reduce the adverse reactions of analgesic and sedative drugs compared with remifentanil combined with propofol.

From January 1, 2023 to January 1, 2024, the clinical study of the patients (60 cases) enrolled in the first phase was completed as expected in the study protocol. Stage objective: to count the relevant detection indicators of the two groups of patients, analyze and compare whether there is a difference between the primary endpoint and the secondary observation endpoint, and write a research paper and a mid-term summary.

From January 1, 2024 to January 1, 2025, the clinical study of patients (60 cases) enrolled in the second phase was completed according to the research protocol. Stage objective: to count the relevant detection indicators of the two groups of patients, analyze and compare whether there is a difference between the primary endpoint and the secondary observation endpoint, and write a research paper and a conclusion report.

Publication form of research results: 1-2 academic papers published in domestic or international journals.

ELIGIBILITY:
Inclusion Criteria:

1. Adults (aged 18-75 years)
2. Septic shock patients with invasive mechanical ventilation
3. Use norepinephrine (the only vasoactive drug) to maintain the target map ≥ 65 mmHg
4. BMI 18.5-23.9kg/m2

Exclusion Criteria:

1. Pregnant or lactating women;
2. Patients allergic to planned drugs;
3. Hypertension patients with poor control;
4. Patients with mental illness, chronic pain, seizures, elevated intracranial pressure, severe ischemic heart disease, and bronchial asthma;
5. Patients included in other trial items;
6. Other reasons that the researcher considers unsuitable to participate in this study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Norepinephrine dosage in two groups | 2 years
  mg/kg

SECONDARY OUTCOMES:
Time of mechanical ventilation | During hospitalization, an average of 4 days
  day
The incidence of intestinal dysfunction | 2 years
  percent

REFERENCES:
- [Derived] Li Y, Li H, Zhang F, Chen Y, Zhang D. Effects of Esketamine Versus Remifentanil on Hemodynamics and Prognosis in Patients with Septic Shock Receiving Invasive Mechanical Ventilation: A Randomized Controlled Trial. Drug Des Devel Ther. 2025 May 21;19:4139-4149. doi: 10.2147/DDDT.S520252. eCollection 2025. PMID 40416798